CLINICAL TRIAL: NCT02433548
Title: Fascia Iliaca Block in the Emergency Department for Analgesia After Femoral Neck Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, PD Dr Eric Albrecht, MD, MER, DESA, Program Director, Regional Anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 318/14
Record Dates: First submitted 2014-10-20; First posted 2015-05-05 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Femoral Neck Fracture
Keywords: Analgesia; Emergency medicine; Anesthesia, Regional
MeSH Terms: conditions — Femoral Neck Fractures; Agnosia | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fascia iliaca block (Experimental): Fascia iliaca block (Injection of 30 mLs of bupivacaine 0.5% with epinephrine 5 mcg/mL below the fascia iliaca, Carbostesin®)
  Interventions: Procedure: Fascia iliaca block
- Sham injection (Sham Comparator): No fascia iliaca block (Sham injection = Subcutaneous injection of 5 cc of normal saline, no intervention)
  Interventions: Procedure: Sham injection

INTERVENTIONS:
Procedure: Fascia iliaca block — injection of 30 mLs below the fascia iliaca
  Arms: Fascia iliaca block
Procedure: Sham injection — subcutaneous of 5 cc of normal saline
  Arms: Sham injection

SUMMARY:
Femoral neck fracture is very common in the elderly and can produce severe to moderate pain. As this pathology is not life-threatening, waiting time in the emergency department may be prolonged due to the high number of unforeseen cases with patients remaining in pain.

Fascia iliaca block consists of injecting local anaesthetics below the fascia iliaca, resulting in the anaesthesia of the femoral, the lateral cutaneous and the obturator nerves, with effective analgesia.

DETAILED DESCRIPTION:
The objective of this trial is to compare the fascia iliaca block with a sham injection on patients arriving in the emergency department with a femoral neck fracture.

The fascia iliaca block will be performed with an anatomical landmark technique and a volume of 30 mLs of bupivacaine 0.5% with epinephrine 5 mcg/mL will be injected.

ELIGIBILITY:
Inclusion Criteria:

- patients with femoral neck fracture in the emergency department

Exclusion Criteria:

* presence of demencia
* body weight less than 40kg
* presence of a cancer or patients receiving chemotherapy
* allergy to local anaesthetics

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain scores at rest | 45 minutes after the injection

SECONDARY OUTCOMES:
Pain scores at rest | 60 min, 4h, 8h, 12h, 24h after the injection
Pain scores on movement | 60 min, 4h, 8h, 12h, 24h after the injection
Morphine consumption | 60 min, 4h, 8h, 12h, 24h after the injection
Length of stay | up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- CHUVaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- [Derived] Pasquier M, Taffe P, Hugli O, Borens O, Kirkham KR, Albrecht E. Fascia iliaca block in the emergency department for hip fracture: a randomized, controlled, double-blind trial. BMC Geriatr. 2019 Jul 1;19(1):180. doi: 10.1186/s12877-019-1193-0. PMID 31262265